CLINICAL TRIAL: NCT06374940
Title: The Comparison of Surgical Outcomes to Conventional Hysterectomy and Manipulator-assisted Abdominal Hysterectomy
Brief Title: Surgical Outcomes of Conventional Hysterectomy or Manipulator-assisted Abdominal Hysterectomy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, pınar birol ilter, Specialist of obstetrics and gynecology, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Lütfi Kırdar City Hospital
Record Dates: First submitted 2024-04-16; First posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Gynecologic Disease
Keywords: Hysterectomy, Manipulator-assisted abdominal hysterectomy
MeSH Terms: conditions — Genital Diseases, Female

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- conventional abdominal hysterectomy (No Intervention): The surgical technique of conventional abdominal hysterectomy was described in the literature.
- Manipulator-assisted Abdominal Hysterectomy (Other): In manipulator-assisted abdominal hysterectomy tecnique, a uterine manipulator (SecuFix ® , Richard Wolf) was inserted into the cervix. Conventional hysterectomy steps were performed until the vaginal colpotomy incision. A circular colpotomy incision was made directly over the manipulator silicone cup using a monopolar cautery set at 30W cutting mode without interfering with the cardinal ligament or sacrouterine ligament. The vaginal cuff was sutured using polyglactin 910 (no:1) as a single layer running suture.
  Interventions: Procedure: Manipulator-assisted Abdominal Hysterectomy

INTERVENTIONS:
Procedure: Manipulator-assisted Abdominal Hysterectomy — Manipulator-assisted Abdominal Hysterectomy
  Arms: Manipulator-assisted Abdominal Hysterectomy

SUMMARY:
Objective: The comparison of surgical outcomes conventional hysterectomy and manipulator-assisted hysterectomy

Study design: Prospective randomized controlled trial. Allocation to either group occurred via computer-generated random numbers. Sequentially numbered, opaque envelopes were prepared according to randomization. The patients were unaware of whether they would undergo a conventional hysterectomy or manipulator-assisted abdominal hysterectomy for their surgical procedure. The research coordinator unveiled group assignments upon individual patient recruitment by opening the corresponding envelope.

Study population: Inclusion criteria were patients aged 40-70 years who underwent hysterectomy for benign gynecological indications.

Primary outcomes: (1) Operation Time.

Secondary outcomes: (1) Postoperative early pain (Visual Analog Score (VAS) at 6th and 24th hours of the surgery) (2) intraoperative complications, (3) postoperative complications

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria were patients aged 40-70 years who underwent hysterectomy for benign gynecological indications

Exclusion Criteria:

* Exclusion criteria were patients with additional procedures such as urogynecologic procedures, history of abdominal surgery with midline incision, patients with suspected gynecologic malignancy, endometriosis, tubo-ovarian abscess, pelvic organ prolapse, or those who refused to participate in the study and whose medical records could not be obtained.

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2024-05-17 (Estimated); Study Completion 2024-05-18 (Estimated)

PRIMARY OUTCOMES:
Duration of the surgical procedure | intraoperative
  The surgical operative time was defined as the time from incision to completion of wound closure, also known as 'cut-to-close' time. In the manipulator-assisted abdominal hysterectomy group, the time of uterine manipulator placement was added to the operation time

SECONDARY OUTCOMES:
Postoperative pain at 6th hours | At the 6th hours after the surgical procedure
  Postoperative pain scores will be measured with using Visual Analogue Score (VAS) as self-reported by the participating women. The VAS scores range from 0= no pain to 10= worst imaginable pain.
Postoperative pain at 24th hours | At the 24th hours after the surgical procedure
  postoperative pain scores will be measured with using Visual Analogue Score (VAS) as self-reported by the participating women. The VAS scores range from 0= no pain to 10= worst imaginable pain.
intraoperative complications | Intraoperative
  Any minor and major (e.g., bowel injury, bleeding>300cc, major vessel injury) complications that occur during the surgery
Postoperative complications | Postoperative, in the first month of the surgery
  Any minor and major complications (e.g., bowel injury, haematoma, infection, dyspareunia, vaginal pain, sexual discomfort) that occur in the first month of the surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr.Lütfi Kırdar City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Upon request, after the work is published
Supporting Information: CSR
Time Frame: Upon request, after the work is published, 5 years
Access Criteria: Upon request, after the work is published, 5 years